CLINICAL TRIAL: NCT00194363
Title: The PAL Trial (Physical Activity and Lymphedema)
Brief Title: Strength Training Intervention for Breast Cancer Survivors and the Effects on Lymphedema Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kathryn Schmitz, Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R01CA106851-01 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Lymphedema
Keywords: breast cancer; breast cancer survivors; lymphedema; strength training; breast cancer survivorship
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Strength training — 13 weeks of supervised strength training (twice weekly for 90 minutes per session), 39 weeks of unsupervised strength training (twice weekly for 90 minutes per session)

SUMMARY:
The purpose of the PAL trial is to increase the understanding of the experiences of long-term breast cancer survivors.

Study hypothesis: Strength training will not increase the rate of lymphedema or worsen lymphedema as compared to the non-exercising control participants.

DETAILED DESCRIPTION:
The proposed study will recruit 288 healthy breast cancer survivors (1-15 years post diagnosis, currently free of cancer), in two strata: 144 BrCa survivors with stable lymphedema (defined in section D.2.), and 144 without lymphedema. The women with lymphedema will be 1-15 years post diagnosis. The women without lymphedema will be 1-5 years post diagnosis. The difference in timing is due to the timing of the onset of lymphedema. Because 90% of all lymphedema cases are likely to occur by 5 years post treatment, it would be of greater value to evaluate the safety of strength training for women without lymphedema during the time frame when lymphedema is most likely to develop.

Randomization will be balanced by timing since diagnosis and other factors. Participants will be randomly assigned within lymphedema strata, to the exercise intervention group or the control group. Participants will be recruited in groups (a total of 8 waves) and randomized to either a strength-training group or control group. All outcome measurements will occur at baseline and 12 months later; additionally, all participants will undergo arm volumetry circumference measures, and a subset of arm function tests (range of motion, pain, grip strength) every 3 months.

Protection and safety of all participants All participants will be given access to trained lymphedema specialists throughout study participation, paid for by the study, for evaluation and treatment of lymphedema. Participants without lymphedema will all participate in an educational session led by Dr. Schmitz and co-developed by Ms. Benson and Ms. Oatman to ensure all participants enter the study with a clear understanding of lymphedema.

Each participant with lymphedema will undergo a clinical evaluation to review lymphedema related measures and to assess current management strategies as part of the baseline and 12-month measurement visits. The protocol to standardize the content of these evaluation sessions will be developed in the first twelve months of the study. Participants with lymphedema, who wear a compression garment, will receive two free garments as part of participating in the study. Arm volumes, circumferences, extra-cellular water in the arm and a subset of arm function tests (range of motion, pain, grip strength) will be monitored quarterly in all participants and monthly in treatment group participants. All participants will be encouraged to request more frequent arm volumetry and/or circumferences and/or extra-cellular water in the arm measures if they believe they have had or are concerned about a change of symptoms. Any participant, regardless of group assignment, who experiences the onset or a flare-up of lymphedema will be seen by a trained lymphedema specialist for evaluation and treatment, paid for by the study. Clinical experiences of Ms. Oatman and Ms. Benson suggest that 10% of the participants with lymphedema will experience a flare-up over 12 months of participation.

For purposes of this study, a flare-up will be defined as a 5% increase in inter-limb discrepancy in volume or circumference at the point of greatest visible difference.as persistent pain/achiness/fullness (in the trunk and/or arm), persistent puffiness (visible), or change of color that does not resolve within three days of rest, and that requires 5 or more days of combined decongestive therapy to resolve. Further, for the purposes of this study, onset of lymphedema will be defined as follows: among women not diagnosed with lymphedema prior to study entry, a > 10% inter-limb discrepancy in volume or circumference a the point of greatest visible difference OR swelling or obscuration of anatomic architecture on close inspection OR pitting edema. as a 2 cm or 200 ml or greater difference between the arm treated for breast cancer compared to the unaffected arm in a woman not diagnosed with lymphedema prior to study entry. By these actions and the careful training of the fitness trainers, we will monitor all participants carefully with regard to onset or worsening of lymphedema symptoms.

The intervention group will receive social, behavioral support and research staff contact time to encourage them to increase their activity level to include two weekly strength-training sessions over 12 months. For the first three months, the exercise sessions will be supervised and conducted in small groups of 4, to teach the specifics of the protocol. Thereafter, participants will continue the same exercise protocol on their own or in groups of their choosing. Treatment group participants will be held accountable for completing workouts through exercise logs and reminder calls from research staff. Participants in the treatment group will undergo assessments of arm volumes and circumferences , as well as a subset of arm function tests (range of motion, pain, grip strength) monthly.

The control group will undergo all outcome measures at baseline and 12 months, and a few measures at 3 and 6 months. The outcome measures include assessments of arm circumferences, extra-cellular water in the arm, and volumetry, as well as a subset of arm function tests (range of motion, pain, grip strength), and will be asked to neither make purposeful changes in diet nor to begin strength training until the final measures are completed 12 months later. After completion of the final measures, control group participants will have the option to participate in the same intervention offered to treatment group participants, including a 1-year membership to the YMCA, Sisters in Shape gym, or Pottruck Health and Fitness Center.

ELIGIBILITY:
Inclusion Criteria:

* Women without lymphedema must be 1-5 years post breast cancer diagnosis
* Women with lymphedema must be 1-15 years post breast cancer diagnosis
* Women with lymphedema must have stable lymphedema. ONE of the following:

  * 0-40>10% girth volume difference between the affected and non- affected limb for a non-dominant arm
  * 6-40% girth volume difference between the affected and non- affected limb for a dominant arm inter-limb discrepancy in volume or circumference at the point of greatest visible difference OR swelling or obscuration of anatomic architecture upon close inspection OR pitting edema.

    * 2 cm circumference difference
  * A prior clinical diagnosis of lymphedema and having had any prior intensive lymphedema therapy on the affected arm

As well as ALL of the following four conditions:

* Women with Lymphedema must have ALL of the following:

  * No recorded arm girth change of 15% or greater within the three months.
  * No more than one lymphedema related infection requiring antibiotics within the past 3 months.
  * Participation in all Activities of Daily Living (ADLs) without lymphedema exacerbation for the past 3 months.

Exclusion Criteria:

* For ALL participants (with and without lymphedema)

  * No medical conditions or medications that would prohibit participation in an exercise program or would negatively impact our ability to test our primary aims
  * Not morbidly obese (body mass index >50 kg/m2)
  * No plans for additional (e.g. reconstructive) surgery during the study period
  * No bilateral breast cancers (because this prohibits our ability to assess the primary outcome of interest)
  * No strength training or other upper body resistive exercise within the past year
  * Not planning to move away from the area over the next year
  * Not pregnant or lactating or planning to become pregnant during the study
  * Among women who have given birth: at least 6 months post pregnancy and at least 3 months post lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2005-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Specific aim 1: To determine whether there are any changes in lymphedema in breast cancer survivors who participate in a one-year randomized exercise intervention of twice-weekly strength training, as compared to a non-exercising group. | 1 year

SECONDARY OUTCOMES:
Secondary aim 1: To assess changes in physical functioning of the arms, as measured by tests of range of motion, coordination, pain, and strength that may result from strength training. | 1 year
Secondary aim 2: To assess changes in body composition that may occur from strength training. | 1 year
Secondary aim 3: To assess self-reported changes in health related quality of life, sleep, fatigue, self-esteem, optimism, life satisfaction, sexual function, body image, social support, and general quality of life. | 1 year
Secondary aim 4: To assess changes in psychosocial mediators of exercise behavior, as well as achievement of outcome expectancies that may occur from participation in strength training. | 1 year
Secondary aim 5: To assess changes in biomarkers related to breast cancer, among the participants who start the study with a BMI over 25. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schmitz, PhD, MPH, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Cancer Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Zhang X, Brown JC, Paskett ED, Zemel BS, Cheville AL, Schmitz KH. Changes in arm tissue composition with slowly progressive weight-lifting among women with breast cancer-related lymphedema. Breast Cancer Res Treat. 2017 Jul;164(1):79-88. doi: 10.1007/s10549-017-4221-9. Epub 2017 Apr 8. PMID 28391397
- [Derived] Rogers BH, Brown JC, Gater DR, Schmitz KH. Association Between Maximal Bench Press Strength and Isometric Handgrip Strength Among Breast Cancer Survivors. Arch Phys Med Rehabil. 2017 Feb;98(2):264-269. doi: 10.1016/j.apmr.2016.07.017. Epub 2016 Aug 16. PMID 27543047
- [Derived] Brown JC, Schmitz KH. Weight Lifting and Physical Function Among Survivors of Breast Cancer: A Post Hoc Analysis of a Randomized Controlled Trial. J Clin Oncol. 2015 Jul 1;33(19):2184-9. doi: 10.1200/JCO.2014.57.7395. Epub 2015 May 11. PMID 25964257
- [Derived] Brown JC, Troxel AB, Schmitz KH. Safety of weightlifting among women with or at risk for breast cancer-related lymphedema: musculoskeletal injuries and health care use in a weightlifting rehabilitation trial. Oncologist. 2012;17(8):1120-8. doi: 10.1634/theoncologist.2012-0035. Epub 2012 Jul 2. PMID 22752068
- [Derived] Schmitz KH, Ahmed RL, Troxel AB, Cheville A, Lewis-Grant L, Smith R, Bryan CJ, Williams-Smith CT, Chittams J. Weight lifting for women at risk for breast cancer-related lymphedema: a randomized trial. JAMA. 2010 Dec 22;304(24):2699-705. doi: 10.1001/jama.2010.1837. Epub 2010 Dec 8. PMID 21148134
- [Derived] Schmitz KH, Ahmed RL, Troxel A, Cheville A, Smith R, Lewis-Grant L, Bryan CJ, Williams-Smith CT, Greene QP. Weight lifting in women with breast-cancer-related lymphedema. N Engl J Med. 2009 Aug 13;361(7):664-73. doi: 10.1056/NEJMoa0810118. PMID 19675330